CLINICAL TRIAL: NCT03121274
Title: Early Versus Delayed Pushing in the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 166
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early pushing during vaginal delivery (Active Comparator): patients are allowed to push within one hour after full cervical dilatation whether the vertex was visible or not
  Interventions: Procedure: vaginal delivery
- Delayed pushingduring vaginal delivery (Active Comparator): patients here are asked not to push for maximum of 3 hours or start pushing when the vertex was visible
  Interventions: Procedure: vaginal delivery

INTERVENTIONS:
Procedure: vaginal delivery — vaginal delivery is carried by an expert obstetrician and the need for forceps or ventose is recorded

SUMMARY:
Nulliparous women in spontaneous or induced labour with term singleton pregnancy are randomized into two groups first group (early pushing) in this group patients were allowed to push within one hour after full cervical dilatation whether the vertex was visible or not. Second group (delayed pushing) patients here were asked not to push for maximum of 3 hours or start pushing when the vertex was visible.

DETAILED DESCRIPTION:
Nulliparous women in spontaneous or induced labour with term singleton pregnancy are randomized into two groups first group (early pushing) in this group patients were allowed to push within one hour after full cervical dilatation whether the vertex was visible or not. Second group (delayed pushing) patients here were asked not to push for maximum of 3 hours or start pushing when the vertex was visible.

Oxytocin was allowed in both group and fetus was monitored with CTG.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Gestational age 36 to 40 weeks
* singleton pregnancy

Exclusion Criteria:

* women indicated for cesarean section
* Medical complications of pregnancy as hypertensive disorders or Diabetes Mellitus
* Fetal distress
* Epidural anaesthesia

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 184 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
successful vaginal delivery | within 3 hours from full cervical dilatation
  success of vaginal delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided